CLINICAL TRIAL: NCT00647296
Title: A 2-Part, Randomized, Double-Blind, Safety and Tolerability Study Evaluating KNS-760704 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Safety and Tolerability Study of KNS-760704 in Amyotrophic Lateral Sclerosis (ALS)
Acronym: CL201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Knopp Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KNS-760704-CL201
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Amyotrophic Lateral Sclerosis; Lou Gehrig; Lou Gehrig's; Lou Gehrig's disease; Motor Neuron Disease; Nervous System Diseases; KNS-760704; BIIB050
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Nervous System Diseases | interventions — Dexpramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo during Part 1 and Part 2 placebo washout.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: Placebo or Dexpramipexole (Placebo Comparator): During Part 1, subjects received twice daily doses of dexpramipexole (50 mg/day, 150 mg/day, or 300 mg/day) or matching placebo for approximately 12 weeks.
  Interventions: Drug: Placebo; Drug: Dexpramipexole 50 mg/day; Drug: Dexpramipexole 150 mg/day; Drug: Dexpramipexole 300 mg/day
- Part 2: Placebo washout (Experimental): At the beginning of Part 2, subjects received twice daily doses of placebo for approximately 4 weeks.
  Interventions: Drug: Placebo
- Part 2: Dexpramipexole (Experimental): Following the Part 2 placebo washout, subjects received dexpramipexole (50 mg/day or 300 mg/day), subjects received twice daily doses of placebo for up to 18 months.
  Interventions: Drug: Dexpramipexole 50 mg/day; Drug: Dexpramipexole 300 mg/day

INTERVENTIONS:
Drug: Placebo — Placebo: 2 tablets taken orally twice daily
  Arms: Part 1: Placebo or Dexpramipexole; Part 2: Placebo washout
Drug: Dexpramipexole 50 mg/day — Dexpramipexole: 2 x 12.5 mg tablets taken orally twice daily
  Other Names: KNS-760704; BIIB050
  Arms: Part 1: Placebo or Dexpramipexole; Part 2: Dexpramipexole
Drug: Dexpramipexole 150 mg/day — Dexpramipexole: 2 x 37.5 mg tablets taken orally twice daily
  Other Names: KNS-760704; BIIB050
  Arms: Part 1: Placebo or Dexpramipexole
Drug: Dexpramipexole 300 mg/day — Dexpramipexole: 2 x 75 mg tablets taken orally twice daily
  Other Names: KNS-760704; BIIB050
  Arms: Part 1: Placebo or Dexpramipexole; Part 2: Dexpramipexole

SUMMARY:
This was a 2-part study of dexpramipexole in patients with ALS.

Part 1 was a randomized, placebo-controlled, multi-center study to evaluate the safety, tolerability, and clinical effects of oral administration of 3 dosage levels of dexpramipexole vs. placebo for 12 weeks.

Part 2 was a randomized, double-blind, 2-arm, parallel group, extension study evaluating the safety, tolerability, and clinical effects of oral administration of 2 dosage levels of dexpramipexole for up to 72 weeks.

DETAILED DESCRIPTION:
This study was a two-part, multicenter, double-blind study in subjects with ALS to evaluate the safety and tolerability of dexpramipexole treatment, as well as the preliminary effects on measures of clinical function and mortality of dexpramipexole treatment.

In part 1, 102 subjects with ALS were randomized at 20 US sites to receive placebo, dexpramipexole at 50 mg/day; dexpramipexole at 150 mg/day; or dexpramipexole at 300 mg/day for 12 weeks. Participants who completed Part 1 were eligible to enroll into Part 2.

Part 2 was a randomized, double-blind, 2-arm, parallel-group, extension study evaluating the longer-term safety, tolerability, and clinical effects of oral administration of 2 dosage levels of dexpramipexole. In part 2, following a 4-week, placebo washout, continuing subjects received dexpramipexole at 50 mg/day or 300 mg/day as double-blind treatment for up to 72 additional weeks (Part 2 duration was up to a total of 76 weeks, including the 4 week placebo portion).

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of familial or sporadic ALS, defined as meeting the possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS according to the World Federation of Neurology El Escorial criteria
* Patients with ALS symptom onset < 24 months from randomization
* Patients with upright vital capacity (VC) > 65% of predicted for age, height, and gender

Exclusion Criteria:

* Patients in whom causes of neuromuscular weakness other than ALS have not been excluded
* Patients without clinical evidence of upper motor neuron dysfunction
* Patients with clinically suspected ALS according to the World Federation of Neurology El Escorial criteria
* Patients with prior exposure to KNS-760704 or the R(+) enantiomer of pramipexole (i.e., R(+)-pramipexole)
* Patients taking other investigational agents (including lithium) within 30 days of randomization or during the study

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2008-04-09 (Actual); Primary Completion 2009-07-31 (Actual); Study Completion 2009-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCLA, Dept. of Neurology - Neuromuscular/ALS Research Center, Los Angeles, California
  - The Forbes Norris MDA/ALS Research Center, San Francisco, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusettes General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Bryan LGH Medical Center East, Lincoln, Nebraska
  - Columbia University, Lou Gehrig MDA/ALS Research Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Oregon Health Sciences University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College Of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Sciences Center of San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Cudkowicz M, Bozik ME, Ingersoll EW, Miller R, Mitsumoto H, Shefner J, Moore DH, Schoenfeld D, Mather JL, Archibald D, Sullivan M, Amburgey C, Moritz J, Gribkoff VK. The effects of dexpramipexole (KNS-760704) in individuals with amyotrophic lateral sclerosis. Nat Med. 2011 Nov 20;17(12):1652-6. doi: 10.1038/nm.2579. PMID 22101764

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for the study across 20 recruiting centers US between 09 April 2008 and 26 January 2009 in medical centers located the USA.
Pre-assignment Details: Study conducted in 2 parts: When the first 12 weeks (Part 1) was completed, eligible continuing subjects entered a 4 week placebo washout before being re-randomized to receive either 50 mg/day dexpramipexole or 300 mg/day dexpramipexole for up to 72 additional weeks.
Groups:
- Placebo Twice Daily: Placebo (PBO) BID (twice daily)
- 50 mg/Day Dexpramipexole: dexpramipexole 25 mg BID (twice daily)
- 150 mg/Day Dexpramipexole: dexpramipexole 75 mg BID (twice daily)
- 300 mg/Day Dexpramipexole: dexpramipexole 150 mg BID (twice daily)
Period: Part 1: 12-week Double-Blind Treatment
Arm/Group | Placebo Twice Daily | 50 mg/Day Dexpramipexole | 150 mg/Day Dexpramipexole | 300 mg/Day Dexpramipexole
Started | 27 | 23 | 26 | 26
Completed | 26 | 22 | 26 | 24
Not Completed | 1 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0
Period: Part 2: 4-week Placebo Washout
Arm/Group | Placebo Twice Daily | 50 mg/Day Dexpramipexole | 150 mg/Day Dexpramipexole | 300 mg/Day Dexpramipexole
Started | 97 | 0 | 0 | 0
Completed | 92 | 0 | 0 | 0
Not Completed | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Death | 3 | 0 | 0 | 0
Period: Part 2: 76-week Double-Blind Treatment
Arm/Group | Placebo Twice Daily | 50 mg/Day Dexpramipexole | 150 mg/Day Dexpramipexole | 300 mg/Day Dexpramipexole
Started | 0 | 48 | 0 | 44
Completed | 0 | 33 | 0 | 30
Not Completed | 0 | 15 | 0 | 14
Not completed — Withdrawal by Subject | 0 | 5 | 0 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Death | 0 | 7 | 0 | 5
Not completed — Inability to attend study visits in person | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: all patients who signed an informed consent and were screened for the study, whether randomized or not
Groups:
- Placebo: PBO BID for 12 weeks
- 50 mg/Day: 25 mg BID for 12 weeks
- 150 mg/Day: 75 mg BID for 12 weeks
- 300 mg/Day: 150 mg BID for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | 50 mg/Day | 150 mg/Day | 300 mg/Day | Total
Number analyzed (Participants) | 27 | 23 | 26 | 26 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (9.07) | 58.1 (10.20) | 56.01 (11.03) | 58.2 (10.96) | 57.0 (10.25)
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 7 | 6 | 6 | 8 | 27
  50 to 65 years | 16 | 10 | 17 | 11 | 54
  > 65 years | 4 | 7 | 3 | 7 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 18 | 19 | 65
  Male | 13 | 9 | 8 | 7 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 4 | 2 | 7
  Not Hispanic or Latino | 24 | 22 | 21 | 24 | 91
  Unknown or Not Reported | 2 | 1 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 1 | 4
  White | 25 | 21 | 25 | 24 | 95
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Height [Mean (Standard Deviation); unit: cm] | 170.28 (10.349) | 170.34 (8.209) | 172.22 (12.591) | 174.98 (9.932) | 171.99 (10.471)
Weight [Mean (Standard Deviation); unit: kg] | 74.7 (15.83) | 78.2 (19.89) | 77.4 (18.73) | 82.1 (14.35) | 78.1 (17.18)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 25.66 (3.934) | 26.86 (6.369) | 25.78 (4.492) | 26.81 (4.189) | 26.27 (4.752)

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Hematology Results by Treatment Group
Description: Number of Participants with Potentially Clinically Significant Hematology Results by Treatment Group. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per laboratory test.
Time Frame: 12 weeks
Population: Safety Population: Data from all enrolled subjects who were randomized in Part 1 and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 50 mg/Day: 25 mg dexpramipexole BID for 12 weeks
- 150 mg/Day: 75 mg dexpramipexole BID for 12 weeks
- 300 mg/Day: 150 mg dexpramipexole BID for 12 weeks
Arm/Group | Placebo | 50 mg/Day | 150 mg/Day | 300 mg/Day
Number analyzed (Participants) | 27 | 23 | 26 | 26
Participants
  White Blood Cell Count (x10^3/uL) < 2000/uL | 0 | 0 | 0 | 0
  Neutrophils (x10^3/uL) < 1000/uL | 0 | 0 | 0 | 0
  Eosinophils (x10^3/uL) > 5000/uL | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) < 8 g/dL | 0 | 0 | 0 | 0
  Platelets (x10^3/uL) < 50,000/uL | 0 | 0 | 0 | 0

2. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Blood Chemistry Results by Treatment Group
Description: Number of Participants with Potentially Clinically Significant Blood Chemistry Results by Treatment Group. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per laboratory test.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/Day | 150 mg/Day | 300 mg/Day
Number analyzed (Participants) | 27 | 23 | 26 | 26
Participants
  Creatine Kinase (U/L) >= 10xULN | 0 | 0 | 0 | 1
  Total Bilirubin (mg/dL) > 1.5xULN | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L) > 3xULN | 0 | 0 | 0 | 2
  AST (SGOT) (U/L) > 3xULN | 0 | 0 | 0 | 1
  Alkaline Phosphatase (U/L) > 1.5xULN | 0 | 0 | 0 | 1
  BUN (mg/dL) > 5xULN | 0 | 0 | 0 | 0
  Creatinine (mg/dL) > 3xULN | 0 | 0 | 0 | 0
  Sodium (mEq/L) low < 123 mEq/L | 0 | 0 | 0 | 0
  Sodium (mEq/L) high > 157 mEq/L | 0 | 0 | 0 | 0
  Potassium (mEq/L) Low < 2.5 mEq/L | 0 | 0 | 0 | 0
  Potassium (mEq/L) High > 6.5 mEq/L | 0 | 0 | 0 | 0
  Glucose (mg/dL) Low < 40 mg/dL | 0 | 0 | 0 | 0
  Glucose (mg/dL) High > 250 mg/dL | 1 | 0 | 0 | 0
  Calcium (mg/dL) Low < 7 mg/dL | 0 | 0 | 0 | 0
  Calcium (mg/dL) High > 12.5 mg/dL | 0 | 0 | 0 | 0

3. Primary Outcome: Part 1: Number of Participants With Treatment Emergent Potentially Clinically Significant Electrocardiogram (ECG) Findings by Treatment Group
Description: Number of Participants with Treatment Emergent Potentially Clinically Significant Electrocardiogram (ECG) Findings by Treatment Group. Percentages are based on the number of patients with at least one non-missing post-baseline value in each treatment group.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/Day | 150 mg/Day | 300 mg/Day
Number analyzed (Participants) | 27 | 23 | 26 | 26
Participants
  Rhythm Sinus Tachycardia > 120 bpm | 0 | 0 | 0 | 0
  Rhythm Sinus Bradycardia < 40 bpm | 0 | 0 | 0 | 0
  Rhythm Sinus Block/Sinus Arrest | 0 | 0 | 0 | 0
  Rhythm Junctional Rhythm | 0 | 0 | 0 | 0
  Rhythm Atrial Flutter | 0 | 0 | 0 | 0
  Rhythm Atrial Fibrillation | 0 | 0 | 0 | 1
  Rhythm Supraventricular | 0 | 0 | 0 | 0
  Rhythm Tachycardia > 100 bpm | 0 | 0 | 0 | 0
  Rhythm Torsades de Pointes | 0 | 0 | 0 | 0
  Rhythm Other Ventricular Rhythm | 0 | 0 | 0 | 0
  Conduction 1st Degree A-V Block | 0 | 1 | 0 | 0
  Conduction 2nd Degree A-V Block | 0 | 0 | 0 | 0
  Conduction 3rd Degree A-V Block | 0 | 0 | 0 | 0
  Conduction Left Bundle Branch Block | 0 | 0 | 0 | 0
  Conduction Right Bundle Branch Block | 0 | 0 | 1 | 0
  Conduction Pre-excitation (PR < 120 msec) | 0 | 0 | 0 | 0
  Conduction Prolonged QTcB | 3 | 3 | 1 | 3
  Conduction Prolonged QTcF | 0 | 0 | 0 | 1
  Myocardial Ischemia/Infarction Myocardial Ischemia | 0 | 1 | 0 | 0
  Myocardial Ischemia/Infarction Possible Myocardial Ischemia | 0 | 0 | 0 | 1
  Myocardial Ischemia/Infarction Old Myocardial Infarction | 1 | 1 | 0 | 0
  Myocardial Ischemia/Infarction Acute or Subacute Myocardial Infarction | 0 | 0 | 0 | 0
  Myocardial Ischemia/Infarction Possible Myocardial Infarction | 3 | 2 | 3 | 0
  U Wave Abnormal U wave present | 0 | 0 | 0 | 0

4. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Vital Sign Measurements by Treatment Group
Description: Number of Participants with Potentially Clinically Significant Vital Sign Measurements by Treatment Group. Percentages are based on the number of patients with at least one non-missing post-baseline value in each treatment group.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/Day | 150 mg/Day | 300 mg/Day
Number analyzed (Participants) | 27 | 23 | 26 | 26
Participants
  Systolic Blood Pressure Increase of > 20 mmHg from baseline and >= 180mmHg | 0 | 2 | 0 | 0
  Systolic Blood Pressure Decrease of < -20 mmHg from baseline and <= 90 mmHg | 2 | 0 | 0 | 0
  Diastolic Blood Pressure Increase of > 15 mmHg from baseline and >= 105 mmHg | 0 | 1 | 0 | 0
  Diastolic Blood Pressure Decrease of < -15 mmHg from baseline and <= 50 mmHg | 1 | 1 | 0 | 0
  Pulse Increase of > 15 bpm from baseline and >= 120 | 0 | 1 | 0 | 0
  Pulse Decrease of < -15 bpm from baseline and <= 50 | 0 | 0 | 0 | 1
  Body Weight Increase of > 7% lbs from baseline | 0 | 0 | 0 | 0
  Body Weight Decrease of < -7% lbs from baseline | 3 | 2 | 0 | 1

5. Secondary Outcome: Part 1: Slope of ALSFRS-R (ALS Functional Rating Scale With Respiratory Component) From Baseline to Week 12 by Treatment Group
Description: The ALSFRS-R (ALS functional rating scale with respiratory component) is a validated scale which measures 4 functional domains, comprising respiratory function, bulbar function, gross motor skills, and fine motor skills. There are a total of 12 questions, each scored from 0 to 4 for a total possible score of 48, with higher scores representing better function. Slope is calculated using a linear mixed effects model with x-axis time in months and y-axis ALSFRS-R score. Units for slope are change per month in units on the ALSFRS-R scale.
Time Frame: 12 weeks
Population: Randomized subjects who had at least 1 post-baseline clinical status evaluation within 7 days of discontinuing study drug
Measure: Least Squares Mean (95% Confidence Interval); unit: slope
Groups:
- Placebo: Two matching PBO tablets taken orally twice daily for 12 weeks
- Dexpramipexole (50 mg/Day): Two 12.5 mg tablets taken orally twice daily for 12 weeks
- Dexpramipexole (150 mg/Day): Two 37.5 mg tablets taken orally twice daily for 12 weeks
- Dexpramipexole (300 mg/Day): Two 75 mg tablets taken orally twice daily for 12 weeks
Arm/Group | Placebo | Dexpramipexole (50 mg/Day) | Dexpramipexole (150 mg/Day) | Dexpramipexole (300 mg/Day)
Number analyzed (Participants) | 27 | 23 | 26 | 26
slope | -1.278 [-1.82 to -0.74] | -1.885 [-2.48 to -1.29] | -1.165 [-1.71 to -0.62] | -0.878 [-1.44 to -0.31]
Statistical Analysis 1: Comparison: Placebo vs Dexpramipexole (50 mg/Day); Test type: Superiority; p = 0.1385, Mixed Models Analysis; Slope = -0.606, 95% CI 2-sided [-1.41 to 0.19], Standard Error of Mean 0.408 — placebo minus active treatment arm, positive direction represents better outcome
Statistical Analysis 2: Comparison: Placebo vs Dexpramipexole (150 mg/Day); Test type: Superiority; p = 0.7718, Mixed Models Analysis; Slope = 0.113, 95% CI 2-sided [-0.65 to 0.88], Standard Error of Mean 0.390 — placebo minus active treatment arm, positive direction represents better outcome
Statistical Analysis 3: Comparison: Placebo vs Dexpramipexole (300 mg/Day); Test type: Superiority; p = 0.3146, Mixed Models Analysis; Slope = 0.401, 95% CI 2-sided [-0.38 to 1.18], Standard Error of Mean 0.397 — placebo minus active treatment arm, positive direction represents better outcome

6. Secondary Outcome: Part 1: Slope of Upright Vital Capacity From Baseline to Week 12 by Treatment Group
Description: Slope of change in Upright Vital Capacity (percent predicted upright vital capacity) from Baseline to Week 12. A negative change/slope indicates clinical worsening. Slope is calculated using a linear mixed effects model with x-axis time in months and y-axis as percent predicted upright vital capacity. Units for slope are change per month in percent predicted upright vital capacity.
Time Frame: 12 weeks
Population: Randomized subjects who had at least 1 post-baseline clinical status evaluation with 7 days of discontinuing study drug
Measure: Least Squares Mean (95% Confidence Interval); unit: slope
Arm/Group | Placebo | Dexpramipexole (50 mg/Day) | Dexpramipexole (150 mg/Day) | Dexpramipexole (300 mg/Day)
Number analyzed (Participants) | 27 | 23 | 26 | 26
slope | -4.398 [-6.42 to -2.38] | -4.003 [-6.23 to -1.77] | -2.389 [-4.44 to -0.34] | -3.947 [-6.07 to -1.82]
Statistical Analysis 1: Comparison: Placebo vs Dexpramipexole (50 mg/Day); Test type: Superiority; p = 0.7973, Mixed Models Analysis; Slope = 0.395, 95% CI 2-sided [-2.61 to 3.40], Standard Error of Mean 1.536 — placebo minus active treatment arm, positive direction represents a better outcome
Statistical Analysis 2: Comparison: Placebo vs Dexpramipexole (150 mg/Day); Test type: Superiority; p = 0.1732, Mixed Models Analysis; Slope = 2.009, 95% CI 2-sided [-0.87 to 4.89], Standard Error of Mean 1.470 — placebo minus active treatment arm, positive direction represents better outcome
Statistical Analysis 3: Comparison: Placebo vs Dexpramipexole (300 mg/Day); Test type: Superiority; p = 0.7635, Mixed Models Analysis; Slope = 0.451, 95% CI 2-sided [-2.48 to 3.39], Standard Error of Mean 1.497 — placebo minus active treatment arm, positive direction represents a better outcome

7. Secondary Outcome: Part 2 Placebo Washout: Number of Participants With Potentially Clinically Significant Hematology
Description: as for outcome 1
Time Frame: 4 weeks
Population: Safety Population: Data from all enrolled subjects who were randomized in Part 1 and received at least 1 dose of study drug during the placebo washout.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Part 2: 4-week placebo washout
Arm/Group | Placebo
Number analyzed (Participants) | 90
Participants
  White Blood Cell Count (x10^3/uL) < 2000/uL | 0
  Neutrophils (x10^3/uL) < 1000/uL | 0
  Eosinophils (x10^3/uL) > 5000/uL | 0
  Hemoglobin (g/dL) < 8 g/dL | 0
  Platelets (x10^3/uL) < 50,000/uL | 0

8. Secondary Outcome: Part 2 Placebo Washout: Number of Participants With Potentially Clinically Significant Blood Chemistry Results
Description: as for outcome 2
Time Frame: 4 weeks
Population: Safety Population: Data from all enrolled subjects who were randomized in Part 2, received at least 1 dose of study drug, and had one post BL evaluation during the placebo washout.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 97
Participants
  Creatine Kinase (U/L) >= 10xULN: number analyzed (Participants) | 89
  Creatine Kinase (U/L) >= 10xULN | 0
  Total Bilirubin (mg/dL) > 1.5xULN: number analyzed (Participants) | 88
  Total Bilirubin (mg/dL) > 1.5xULN | 0
  ALT (SGPT) (U/L) > 3xULN: number analyzed (Participants) | 89
  ALT (SGPT) (U/L) > 3xULN | 0
  AST (SGOT) (U/L) > 3xULN: number analyzed (Participants) | 87
  AST (SGOT) (U/L) > 3xULN | 0
  Alkaline Phosphatase (U/L) > 1.5xULN: number analyzed (Participants) | 90
  Alkaline Phosphatase (U/L) > 1.5xULN | 0
  BUN (mg/dL) > 5xULN: number analyzed (Participants) | 90
  BUN (mg/dL) > 5xULN | 0
  Creatinine (mg/dL) > 3xULN: number analyzed (Participants) | 90
  Creatinine (mg/dL) > 3xULN | 0
  Sodium (mEq/L) low < 123 mEq/L: number analyzed (Participants) | 89
  Sodium (mEq/L) low < 123 mEq/L | 0
  Sodium (mEq/L) high > 157 mEq/L: number analyzed (Participants) | 89
  Sodium (mEq/L) high > 157 mEq/L | 0
  Potassium (mEq/L) Low < 2.5 mEq/L: number analyzed (Participants) | 89
  Potassium (mEq/L) Low < 2.5 mEq/L | 0
  Potassium (mEq/L) High > 6.5 mEq/L: number analyzed (Participants) | 89
  Potassium (mEq/L) High > 6.5 mEq/L | 0
  Glucose (mg/dL) Low < 40 mg/dL: number analyzed (Participants) | 89
  Glucose (mg/dL) Low < 40 mg/dL | 0
  Glucose (mg/dL) High > 250 mg/dL: number analyzed (Participants) | 89
  Glucose (mg/dL) High > 250 mg/dL | 0
  Calcium (mg/dL) Low < 7 mg/dL: number analyzed (Participants) | 90
  Calcium (mg/dL) Low < 7 mg/dL | 0
  Calcium (mg/dL) High > 12.5 mg/dL: number analyzed (Participants) | 90
  Calcium (mg/dL) High > 12.5 mg/dL | 0

9. Secondary Outcome: Part 2 Placebo Washout: Number of Participants With Treatment Emergent Potentially Clinically Significant Electrocardiogram (ECG) Findings
Description: as for outcome 3
Time Frame: 4 weeks
Population: Safety Population: Data from all enrolled subjects who were randomized in Part 1, received at least 1 dose of study drug, and have at least on evaluation post baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 97
Participants
  Rhythm Sinus Tachycardia > 120 bpm: number analyzed (Participants) | 92
  Rhythm Sinus Tachycardia > 120 bpm | 0
  Rhythm Sinus Bradycardia < 40 bpm: number analyzed (Participants) | 92
  Rhythm Sinus Bradycardia < 40 bpm | 0
  Rhythm Sinus Block/Sinus Arrest: number analyzed (Participants) | 92
  Rhythm Sinus Block/Sinus Arrest | 0
  Rhythm Junctional Rhythm: number analyzed (Participants) | 92
  Rhythm Junctional Rhythm | 0
  Rhythm Atrial Flutter: number analyzed (Participants) | 92
  Rhythm Atrial Flutter | 0
  Rhythm Atrial Fibrillation: number analyzed (Participants) | 92
  Rhythm Atrial Fibrillation | 0
  Rhythm Supraventricular: number analyzed (Participants) | 92
  Rhythm Supraventricular | 0
  Rhythm Tachycardia > 100 bpm: number analyzed (Participants) | 92
  Rhythm Tachycardia > 100 bpm | 0
  Rhythm Torsades de Pointes: number analyzed (Participants) | 92
  Rhythm Torsades de Pointes | 0
  Rhythm Other Ventricular Rhythm: number analyzed (Participants) | 92
  Rhythm Other Ventricular Rhythm | 0
  Conduction 1st Degree A-V Block: number analyzed (Participants) | 86
  Conduction 1st Degree A-V Block | 2
  Conduction 2nd Degree A-V Block: number analyzed (Participants) | 86
  Conduction 2nd Degree A-V Block | 0
  Conduction 3rd Degree A-V Block: number analyzed (Participants) | 86
  Conduction 3rd Degree A-V Block | 0
  Conduction Left Bundle Branch Block: number analyzed (Participants) | 86
  Conduction Left Bundle Branch Block | 0
  Conduction Right Bundle Branch Block: number analyzed (Participants) | 86
  Conduction Right Bundle Branch Block | 2
  Conduction Pre-excitation (PR < 120 msec): number analyzed (Participants) | 86
  Conduction Pre-excitation (PR < 120 msec) | 0
  Conduction Prolonged QTcB: number analyzed (Participants) | 86
  Conduction Prolonged QTcB | 4
  Conduction Prolonged QTcF: number analyzed (Participants) | 86
  Conduction Prolonged QTcF | 3
  Myocardial Ischemia/Infarction Myocardial Ischemia: number analyzed (Participants) | 86
  Myocardial Ischemia/Infarction Myocardial Ischemia | 0
  Myocardial Ischemia/Infarction Possible Myocardial Ischemia: number analyzed (Participants) | 86
  Myocardial Ischemia/Infarction Possible Myocardial Ischemia | 2
  Myocardial Ischemia/Infarction Old Myocardial Infarction: number analyzed (Participants) | 86
  Myocardial Ischemia/Infarction Old Myocardial Infarction | 4
  Myocardial Ischemia/Infarction Acute or Subacute Myocardial Infarction: number analyzed (Participants) | 86
  Myocardial Ischemia/Infarction Acute or Subacute Myocardial Infarction | 0
  Myocardial Ischemia/Infarction Possible Myocardial Infarction: number analyzed (Participants) | 86
  Myocardial Ischemia/Infarction Possible Myocardial Infarction | 4
  U Wave Abnormal U wave present: number analyzed (Participants) | 86
  U Wave Abnormal U wave present | 0

10. Secondary Outcome: Part 2 Placebo Washout: Number of Participants With Potentially Clinically Significant Vital Sign Measurements
Description: as for outcome 4
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 97
Participants
  Systolic Blood Pressure Increase of > 20 mmHg from baseline and >= 180mmHg: number analyzed (Participants) | 92
  Systolic Blood Pressure Increase of > 20 mmHg from baseline and >= 180mmHg | 0
  Systolic Blood Pressure Decrease of < -20 mmHg from baseline and <= 90 mmHg: number analyzed (Participants) | 92
  Systolic Blood Pressure Decrease of < -20 mmHg from baseline and <= 90 mmHg | 0
  Diastolic Blood Pressure Increase of > 15 mmHg from baseline and >= 105 mmHg: number analyzed (Participants) | 92
  Diastolic Blood Pressure Increase of > 15 mmHg from baseline and >= 105 mmHg | 2
  Diastolic Blood Pressure Decrease of < -15 mmHg from baseline and <= 50 mmHg: number analyzed (Participants) | 92
  Diastolic Blood Pressure Decrease of < -15 mmHg from baseline and <= 50 mmHg | 0
  Pulse Increase of > 15 bpm from baseline and >= 120: number analyzed (Participants) | 92
  Pulse Increase of > 15 bpm from baseline and >= 120 | 1
  Pulse Decrease of < -15 bpm from baseline and <= 50: number analyzed (Participants) | 92
  Pulse Decrease of < -15 bpm from baseline and <= 50 | 1
  Body Weight Increase of > 7% lbs from baseline: number analyzed (Participants) | 90
  Body Weight Increase of > 7% lbs from baseline | 0
  Body Weight Decrease of < -7% lbs from baseline: number analyzed (Participants) | 90
  Body Weight Decrease of < -7% lbs from baseline | 0

11. Secondary Outcome: Part 2 Placebo Washout: Absolute Change in ALSFRS-R Total Score
Description: The ALSFRS-R (ALS functional rating scale with respiratory component) is a validated scale which measures 4 functional domains, comprising respiratory function, bulbar function, gross motor skills, and fine motor skills. There are a total of 12 questions, each scored from 0 to 4 for a total possible score of 48, with higher scores representing better function.
  Units are points on the ALSFRS-R score as an absolute change from the baseline of the placebo washout to week 4 of the placebo washout.
Time Frame: 4 weeks
Population: Randomized subjects who had at least 1 post-baseline clinical status evaluation with 7 days of discontinuing study drug
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo
Number analyzed (Participants) | 92
units on a scale | -1.2 (0.27)

12. Secondary Outcome: Part 2 Placebo Washout: Absolute Change in Upright Vital Capacity (Percent Predicted) From Baseline to End of Placebo Washout (Week 4)
Description: Absolute change in Upright Vital Capacity From Baseline to Week 4. Units are percent of predicted Upright Vital Capacity. A negative change indicates clinical worsening.
Time Frame: 4 weeks
Population: Randomized subjects who had at least 1 post-baseline clinical status evaluation with 7 days of discontinuing study drug
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo
Number analyzed (Participants) | 89
units on a scale | -3.1 (0.95)

13. Secondary Outcome: Part 2 Double-Blind Treatment: Number of Participants With Potentially Clinically Significant Hematology Results by Treatment Group
Description: Number of Participants with Potentially Clinically Significant Hematology Results by Treatment Group. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per parameter.
Time Frame: up to 76 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/Day | 300 mg/Day
Number analyzed (Participants) | 48 | 44
Participants
  White Blood Cell Count (x10^3/uL) < 2000/uL | 0 | 0
  Neutrophils (x10^3/uL) < 1000/uL | 0 | 0
  Eosinophils (x10^3/uL) > 5000/uL | 0 | 0
  Hemoglobin (g/dL) < 8 g/dL | 0 | 1
  Platelets (x10^3/uL) < 50,000/uL | 0 | 0

14. Secondary Outcome: Part 2 Double-Blind Treatment: Number of Participants With Potentially Clinically Significant Blood Chemistry Results by Treatment Group
Description: Number of Participants with Potentially Clinically Significant Blood Chemistry Results by Treatment Group. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per parameter.
Time Frame: up to 76 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/Day | 300 mg/Day
Number analyzed (Participants) | 48 | 44
Participants
  Creatine Kinase (U/L) >= 10xULN: number analyzed (Participants) | 47 | 44
  Creatine Kinase (U/L) >= 10xULN | 0 | 0
  Total Bilirubin (mg/dL) > 1.5xULN: number analyzed (Participants) | 47 | 44
  Total Bilirubin (mg/dL) > 1.5xULN | 0 | 0
  ALT (SGPT) (U/L) > 3xULN: number analyzed (Participants) | 47 | 44
  ALT (SGPT) (U/L) > 3xULN | 1 | 2
  AST (SGOT) (U/L) > 3xULN: number analyzed (Participants) | 47 | 44
  AST (SGOT) (U/L) > 3xULN | 1 | 0
  Alkaline Phosphatase (U/L) > 1.5xULN: number analyzed (Participants) | 47 | 44
  Alkaline Phosphatase (U/L) > 1.5xULN | 1 | 1
  BUN (mg/dL) > 5xULN: number analyzed (Participants) | 47 | 44
  BUN (mg/dL) > 5xULN | 0 | 0
  Creatinine (mg/dL) > 3xULN: number analyzed (Participants) | 47 | 44
  Creatinine (mg/dL) > 3xULN | 0 | 0
  Sodium (mEq/L) low < 123 mEq/L: number analyzed (Participants) | 47 | 44
  Sodium (mEq/L) low < 123 mEq/L | 0 | 0
  Sodium (mEq/L) high > 157 mEq/L: number analyzed (Participants) | 47 | 44
  Sodium (mEq/L) high > 157 mEq/L | 1 | 0
  Potassium (mEq/L) Low < 2.5 mEq/L: number analyzed (Participants) | 47 | 44
  Potassium (mEq/L) Low < 2.5 mEq/L | 0 | 1
  Potassium (mEq/L) High > 6.5 mEq/L: number analyzed (Participants) | 47 | 44
  Potassium (mEq/L) High > 6.5 mEq/L | 0 | 0
  Glucose (mg/dL) Low < 40 mg/dL: number analyzed (Participants) | 47 | 44
  Glucose (mg/dL) Low < 40 mg/dL | 0 | 0
  Glucose (mg/dL) High > 250 mg/dL: number analyzed (Participants) | 47 | 44
  Glucose (mg/dL) High > 250 mg/dL | 1 | 1
  Calcium (mg/dL) Low < 7 mg/dL: number analyzed (Participants) | 47 | 44
  Calcium (mg/dL) Low < 7 mg/dL | 0 | 1
  Calcium (mg/dL) High > 12.5 mg/dL: number analyzed (Participants) | 47 | 44
  Calcium (mg/dL) High > 12.5 mg/dL | 0 | 0

15. Secondary Outcome: Part 2 Double-Blind Treatment: Number of Participants With Treatment Emergent Potentially Clinically Significant Electrocardiogram (ECG) Findings by Treatment Group
Description: Number of Participants with Treatment Emergent Potentially Clinically Significant Electrocardiogram (ECG) Findings by Treatment Group. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per parameter.
Time Frame: up to 76 weeks
Population: Safety Population: Data from all enrolled subjects who were randomized in Part 2, received at least 1 dose of study drug, and had at least one evaluation post baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/Day | 300 mg/Day
Number analyzed (Participants) | 48 | 44
Participants
  Rhythm Sinus Tachycardia > 120 bpm | 2 | 0
  Rhythm Sinus Bradycardia < 40 bpm | 0 | 0
  Rhythm Sinus Block/Sinus Arrest | 0 | 0
  Rhythm Junctional Rhythm | 0 | 1
  Rhythm Atrial Flutter | 0 | 0
  Rhythm Atrial Fibrillation | 0 | 1
  Rhythm Supraventricular | 0 | 0
  Rhythm Tachycardia > 100 bpm | 0 | 0
  Rhythm Torsades de Pointes | 0 | 0
  Rhythm Other Ventricular Rhythm | 0 | 0
  Conduction 1st Degree A-V Block | 2 | 2
  Conduction 2nd Degree A-V Block | 0 | 0
  Conduction 3rd Degree A-V Block | 0 | 0
  Conduction Left Bundle Branch Block | 0 | 0
  Conduction Right Bundle Branch Block | 1 | 2
  Conduction Pre-excitation (PR < 120 msec) | 0 | 0
  Conduction Prolonged QTcB | 6 | 3
  Conduction Prolonged QTcF | 1 | 1
  Myocardial Ischemia/Infarction Myocardial Ischemia | 0 | 0
  Myocardial Ischemia/Infarction Possible Myocardial Ischemia | 1 | 0
  Myocardial Ischemia/Infarction Old Myocardial Infarction | 3 | 2
  Myocardial Ischemia/Infarction Acute or Subacute Myocardial Infarction | 0 | 0
  Myocardial Ischemia/Infarction Possible Myocardial Infarction | 4 | 2
  U Wave Abnormal U wave present | 0 | 0

16. Secondary Outcome: Part 2 Double-Blind Treatment: Number of Participants With Potentially Clinically Significant Vital Sign Measurements by Treatment Group
Description: Number of Participants with Potentially Clinically Significant Vital Sign Measurements by Treatment Group. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per parameter.
Time Frame: up to 76 weeks
Population: Safety Population: Data from all enrolled subjects who were randomized in Part 1, received at least 1 dose of study drug, and had at least one post baseline evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/Day | 300 mg/Day
Number analyzed (Participants) | 48 | 44
Participants
  Systolic Blood Pressure Increase of > 20 mmHg from baseline and >= 180mmHg | 0 | 0
  Systolic Blood Pressure Decrease of < -20 mmHg from baseline and <= 90 mmHg | 0 | 1
  Diastolic Blood Pressure Increase of > 15 mmHg from baseline and >= 105 mmHg | 2 | 1
  Diastolic Blood Pressure Decrease of < -15 mmHg from baseline and <= 50 mmHg | 3 | 1
  Pulse Increase of > 15 bpm from baseline and >= 120 | 1 | 2
  Pulse Decrease of < -15 bpm from baseline and <= 50 | 0 | 0
  Body Weight Increase of > 7% lbs from baseline: number analyzed (Participants) | 44 | 42
  Body Weight Increase of > 7% lbs from baseline | 1 | 1
  Body Weight Decrease of < -7% lbs from baseline: number analyzed (Participants) | 44 | 42
  Body Weight Decrease of < -7% lbs from baseline | 14 | 16

17. Secondary Outcome: Part 2 Double-Blind Treatment: Slope of the ALSFRS-R (ALS Functional Rating Scale With Respiratory Component) From Baseline to Week 28 by Treatment Group
Description: The ALSFRS-R (ALS functional rating scale with respiratory component) is a validated scale which measures 4 functional domains, comprising respiratory function, bulbar function, gross motor skills, and fine motor skills. There are a total of 12 questions, each scored from 0 to 4 for a total possible score of 48, with higher scores representing better function. Slope is calculated using a linear mixed effects model with x-axis time in months and y-axis ALSFRS-R score. Units for slope are change per month n units on the ALSFRS-R scale.
Time Frame: 28 weeks
Population: Randomized subjects who had at least 1 post-baseline clinical status evaluation with 7 days of discontinuing study drug
Measure: Least Squares Mean (95% Confidence Interval); unit: slope
Arm/Group | Dexpramipexole (50 mg/Day) | Dexpramipexole (300 mg/Day)
Number analyzed (Participants) | 46 | 44
slope | -1.284 [-1.56 to -1.01] | -1.021 [-1.29 to -0.75]
Statistical Analysis 1: Comparison: Dexpramipexole (50 mg/Day) vs Dexpramipexole (300 mg/Day); Test type: Superiority; p = 0.1772, Mixed Models Analysis; Slope = 0.263, 95% CI 2-sided [-0.12 to 0.64], Standard Error of Mean 0.19 — 50 mg/day minus 150 mg/day arm, negative direction represents worse outcome

18. Secondary Outcome: Part 2 Double-Blind Treatment: Slope of Percent Predicted Upright Vital Capacity From Baseline by Treatment Group
Description: Slope of Upright Vital Capacity (percent predicted) through Week 28. A negative change indicates clinical worsening. Slope is calculated using a linear mixed effects model with x-axis time in months and y-axis percent predicted upright vital capacity. Units for slope are change per month in percent predicted upright vital capacity.
Time Frame: Baseline of randomized phase of Part 2 to week 28 of randomized phase of Part 2
Population: Randomized subjects who had at least 1 post-baseline clinical status evaluation with 7 days of discontinuing study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: slope
Arm/Group | Dexpramipexole (50 mg/Day) | Dexpramipexole (300 mg/Day)
Number analyzed (Participants) | 46 | 44
slope | -2.452 [-3.50 to -1.41] | -3.067 [-4.06 to -2.07]
Statistical Analysis 1: Comparison: Dexpramipexole (50 mg/Day) vs Dexpramipexole (300 mg/Day); Test type: Superiority; p = 0.4025, Mixed Models Analysis; Slope = -0.615, 95% CI 2-sided [-2.06 to 0.83], Standard Error of Mean 0.73 — 50 mg/day minus 300 mg/day treatment arm, negative direction represents worse outcome

ADVERSE EVENTS:
Time Frame: Part 1: up to 12 weeks; Part 2 Placebo washout: up to 4 weeks; Part 2 Treatment period: up to 18 months
Groups:
- Part 1: Placebo: Two matching PBO tablets taken orally twice daily for 12 weeks
- Part 1: Dexpramipexole (50 mg/Day): Two 12.5 mg tablets taken orally twice daily for 12 weeks
- Part 1: Dexpramipexole (150 mg/Day): Two 37.5 mg tablets taken orally twice daily for 12 weeks
- Part 1: Dexpramipexole (300 mg/Day): Two 75 mg tablets taken orally twice daily for 12 weeks
- Part 2: Placebo Washout: Two matching PBO tablets taken orally twice daily for 4 weeks
- Part 2: Dexpramipexole (50 mg/Day): Two 12.5 mg tablets taken orally twice daily for up to 18 months
- Part 2: Dexpramipexole (300 mg/Day): Two 75 mg tablets taken orally twice daily for up to 18 months
Arm/Group | Part 1: Placebo | Part 1: Dexpramipexole (50 mg/Day) | Part 1: Dexpramipexole (150 mg/Day) | Part 1: Dexpramipexole (300 mg/Day) | Part 2: Placebo Washout | Part 2: Dexpramipexole (50 mg/Day) | Part 2: Dexpramipexole (300 mg/Day)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/23 | 0/26 | 0/26 | 3/97 | 15/48 | 9/44
Serious Adverse Events (participants affected / at risk) | 0/27 | 2/23 | 0/26 | 3/26 | 5/97 | 14/48 | 12/44
Other Adverse Events (participants affected / at risk) | 25/27 | 19/23 | 25/26 | 23/26 | 46/97 | 46/48 | 41/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=27) | Part 1: Dexpramipexole (50 mg/Day) (N=23) | Part 1: Dexpramipexole (150 mg/Day) (N=26) | Part 1: Dexpramipexole (300 mg/Day) (N=26) | Part 2: Placebo Washout (N=97) | Part 2: Dexpramipexole (50 mg/Day) (N=48) | Part 2: Dexpramipexole (300 mg/Day) (N=44)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
INTESTINAL INFARCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DISEASE PROGRESSION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUDDEN DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CHOKING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=27) | Part 1: Dexpramipexole (50 mg/Day) (N=23) | Part 1: Dexpramipexole (150 mg/Day) (N=26) | Part 1: Dexpramipexole (300 mg/Day) (N=26) | Part 2: Placebo Washout (N=97) | Part 2: Dexpramipexole (50 mg/Day) (N=48) | Part 2: Dexpramipexole (300 mg/Day) (N=44)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 4
Constipation (Gastrointestinal disorders) | 5 | 1 | 3 | 2 | 6 | 8 | 11
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 3 | 2 | 4
Dry Mouth (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 1 | 1 | 7
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 4
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 4 | 4 | 5 | 5
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 8 | 8
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Disease Progression (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 3
Fatigue (General disorders) | 2 | 2 | 0 | 2 | 0 | 1 | 3
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 4
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 4
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 5 | 3
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 6 | 5
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 1 | 1 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 6 | 11 | 7 | 11 | 13 | 11
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 7 | 4 | 5 | 5 | 3 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1 | 0 | 2 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 3 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 0 | 1 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 6 | 5 | 7 | 6 | 7 | 15 | 7
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 1 | 0 | 4 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Dysarthria (Nervous system disorders) | 1 | 2 | 1 | 1 | 0 | 4 | 5
Headache (Nervous system disorders) | 5 | 1 | 3 | 6 | 2 | 5 | 6
Muscle Contractions Involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2
Muscle Spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1
Affect Lability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 6
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 6 | 8
Insomnia (Psychiatric disorders) | 1 | 3 | 1 | 1 | 1 | 0 | 9
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 6 | 2 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3 | 3 | 5 | 6
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other